CLINICAL TRIAL: NCT07072546
Title: Effects of Chitosan and i-PRF on Wound Healing After Palatal Graft Harvesting
Brief Title: Chitosan and i-PRF in Palatal Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Prof., Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chitosan-iPRF
Record Dates: First submitted 2025-07-07; First posted 2025-07-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Free Gingival Graft; Wound Healing; i-PRF; Chitosan
MeSH Terms: interventions — Chitosan; proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control (Other): control group
  Interventions: Procedure: free gingival graft + gelatin sponge
- chitosan (Active Comparator)
  Interventions: Procedure: free gingival graft + chitosan
- chitosan-iprf (Experimental)
  Interventions: Procedure: free gingival graft + chitosan and i-PRF

INTERVENTIONS:
Procedure: free gingival graft + gelatin sponge — Free gingival graft surgery and application of gelatin sponge to the palatal wound
  Arms: control
Procedure: free gingival graft + chitosan — free gingival graft surgery and application of chitosan to the palatal wound
  Arms: chitosan
Procedure: free gingival graft + chitosan and i-PRF — free gingival graft surgery and application of chitosan and i-PRF to the palatal wound
  Arms: chitosan-iprf

SUMMARY:
This study aims to evaluate the effects of chitosan and injectable platelet-rich fibrin (i-PRF) on wound healing at the donor site following free gingival graft (FGG) procedures. The palatal donor area often experiences delayed healing and postoperative discomfort, motivating the search for effective biomaterials to enhance recovery and reduce patient morbidity. Although various approaches have been investigated, the combined application of chitosan and i-PRF has not yet been explored in this context.

The study examines three patient groups treated at the periodontology departments of Çukurova and Biruni University: one with gelatin sponge (control), one with chitosan, and one with chitosan infused with i-PRF. Parameters such as pain (VAS), bleeding, burning sensation, dietary changes, epithelialization (PEHI score), and color match were assessed over a 2-month follow-up.

The findings are expected to provide insights into whether i-PRF-enhanced chitosan offers superior healing outcomes and greater patient comfort compared to conventional methods.

ELIGIBILITY:
Inclusion Criteria:

* Periodontally healthy
* Having good oral hygiene (plaque accumulation <20%)
* Requiring a free gingival graft (FGG) procedure in an area with insufficient keratinized gingiva width (<2 mm)

Exclusion Criteria:

* Having systemic diseases contraindicating surgical procedures,
* Uncontrolled diabetes (HbA1c > 7),
* Being pregnant or breastfeeding,
* Autoimmune and/or inflammatory diseases of the oral cavity,
* Active periodontal disease,
* Smokers (≥ 10 cigarettes per day)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-07-12 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Palatal early healing index | Day 7
  The palatal early healing index (PEHI) measured the following 5 parameters: (1) bleeding on palpation, which was assessed with a damp cotton applicator gently rolled on the wound site; (2) incomplete epithelialization (assessed intraorally by the visual presence or absence of immediate bubble formation after hydrogen peroxide application with sterile gauze on the wound area); (3) presence of redness assessed intraorally; (4) presence of swelling assessed intraorally; and (5) presence of granulation tissue assessed intraorally. Each of the 5 parameters was assessed dichotomously (yes/no).
Palatal early healing index | Day 14
  The palatal early healing index (PEHI) measured the following 5 parameters: (1) bleeding on palpation, which was assessed with a damp cotton applicator gently rolled on the wound site; (2) incomplete epithelialization (assessed intraorally by the visual presence or absence of immediate bubble formation after hydrogen peroxide application with sterile gauze on the wound area); (3) presence of redness assessed intraorally; (4) presence of swelling assessed intraorally; and (5) presence of granulation tissue assessed intraorally. Each of the 5 parameters was assessed dichotomously (yes/no).
Palatal early healing index | Day 28
  The palatal early healing index (PEHI) measured the following 5 parameters: (1) bleeding on palpation, which was assessed with a damp cotton applicator gently rolled on the wound site; (2) incomplete epithelialization (assessed intraorally by the visual presence or absence of immediate bubble formation after hydrogen peroxide application with sterile gauze on the wound area); (3) presence of redness assessed intraorally; (4) presence of swelling assessed intraorally; and (5) presence of granulation tissue assessed intraorally. Each of the 5 parameters was assessed dichotomously (yes/no).
Palatal early healing index | Day 56
  The palatal early healing index (PEHI) measured the following 5 parameters: (1) bleeding on palpation, which was assessed with a damp cotton applicator gently rolled on the wound site; (2) incomplete epithelialization (assessed intraorally by the visual presence or absence of immediate bubble formation after hydrogen peroxide application with sterile gauze on the wound area); (3) presence of redness assessed intraorally; (4) presence of swelling assessed intraorally; and (5) presence of granulation tissue assessed intraorally. Each of the 5 parameters was assessed dichotomously (yes/no).

SECONDARY OUTCOMES:
Palatal Pain score | Day 1
  The degree of pain in the patient's palatal region will be evaluated using visual analogue scale (0-no pain to 10-severe pain).
Palatal Pain score | Day 3
  The degree of pain in the patient's palatal region will be evaluated using visual analogue scale (0-no pain to 10-severe pain).
Palatal Pain score | Day 7
  The degree of pain in the patient's palatal region will be evaluated using visual analogue scale (0-no pain to 10-severe pain).
Palatal Pain score | Day 14
  The degree of pain in the patient's palatal region will be evaluated using visual analogue scale (0-no pain to 10-severe pain).
Palatal Pain score | Day 28
  The degree of pain in the patient's palatal region will be evaluated using visual analogue scale (0-no pain to 10-severe pain).
Palatal Pain score | Day 56
  The degree of pain in the patient's palatal region will be evaluated using visual analogue scale (0-no pain to 10-severe pain).
Use of analgesics and palatal bleeding | Day 1
  Patients will be given a form and asked to record this informations daily.
Difficulty in chewing | Day 7
  The degree of difficulty in chewing in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Difficulty in chewing | Day 14
  The degree of difficulty in chewing in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Difficulty in chewing | Day 28
  The degree of difficulty in chewing in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Difficulty in chewing | Day 56
  The degree of difficulty in chewing in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Use of analgesics and palatal bleeding | Day 2
  Patients will be given a form and asked to record this information daily.
Use of analgesics and palatal bleeding | Day 3
  Patients will be given a form and asked to record this information daily.
Use of analgesics and palatal bleeding | Day 4
  Patients will be given a form and asked to record this information daily.
Use of analgesics and palatal bleeding | Day 5
  Patients will be given a form and asked to record this information daily.
Use of analgesics and palatal bleeding | Day 6
  Patients will be given a form and asked to record this information daily.
Use of analgesics and palatal bleeding | Day 7
  Patients will be given a form and asked to record this information daily.
Graft dimentions | Day 0
  The width, length, and thickness of the palatal graft will be measured using a periodontal probe and recorded.
Color match | Day 14
  The color match at the donor site will be evaluated in comparison with the adjacent palatal area and the contralateral palatal arch by visual analogue scale (0-very bad to 10-excellent).
Color match | Day 28
  The color match at the donor site will be evaluated in comparison with the adjacent palatal area and the contralateral palatal arch by visual analogue scale (0-very bad to 10-excellent).
Color match | Day 56
  The color match at the donor site will be evaluated in comparison with the adjacent palatal area and the contralateral palatal arch by visual analogue scale (0-very bad to 10-excellent).
Burning sensation | Day 1
  The degree of burning sensation in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Burning sensation | Day 3
  The degree of burning sensation in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Burning sensation | Day 7
  The degree of burning sensation in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Burning sensation | Day 14
  The degree of burning sensation in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Burning sensation | Day 28
  The degree of burning sensation in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Burning sensation | Day 56
  The degree of burning sensation in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Changes in dietary habits | Day 1
  The degree of changes in dietary habits in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Changes in dietary habits | Day 3
  The degree of changes in dietary habits in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Changes in dietary habits | Day 7
  The degree of changes in dietary habits in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Changes in dietary habits | Day 14
  The degree of changes in dietary habits in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Changes in dietary habits | Day 28
  The degree of changes in dietary habits in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).
Changes in dietary habits | Day 56
  The degree of changes in dietary habits in the patient's palatal region will be evaluated using visual analogue scale (0-no to 10-severe).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Cukurova University, Adana
  - Biruni University, Istanbul